CLINICAL TRIAL: NCT06849726
Title: Comparison of Standard Epidural and Dural Puncture Epidural Techniques in Labor Analgesia
Brief Title: Epidural vs. Dural Puncture Epidural in Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Burak Omur, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Epidural vs DP epidural
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Labor Pain; Epidural Analgesia
Keywords: Labor Analgesia; Epidural Analgesia; Dural Puncture Epidural
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Epidural Analgesia (Active Comparator): In Group 1, nulliparous women in active labor will receive standard epidural analgesia. After standard monitoring and left lateral positioning, local anesthesia (40 mg of 2% lidocaine) is administered at the L3-L4 or L4-L5 interspace. Using an 18G Tuohy needle and the loss-of-resistance technique, the epidural space is identified, and the epidural catheter is inserted without prior use of a spinal needle. After confirming negative aspiration for CSF or blood, an initial dose of 15 mL of 0.125% bupivacaine with 30 μg fentanyl is administered through the catheter.
  Interventions: Procedure: Standard Epidural Analgesia
- Dural Puncture Epidural (DPE) Analgesia (Active Comparator): In Group 2, nulliparous women in active labor will receive the DPE technique. After identical patient preparation and local anesthetic infiltration at the L3-L4 or L4-L5 interspace, an 18G Tuohy needle is used via the loss-of-resistance method to locate the epidural space. Before inserting the epidural catheter, a 27G spinal needle is introduced through the Tuohy needle to puncture the dura, with the appearance of cerebrospinal fluid (CSF) confirming dural puncture. The spinal needle is then withdrawn without intrathecal drug administration, and the epidural catheter is inserted. Following negative aspiration, the same initial dose of 15 mL of 0.125% bupivacaine with 30 μg fentanyl is administered.
  Interventions: Procedure: Dural Puncture Epidural Analgesia

INTERVENTIONS:
Procedure: Standard Epidural Analgesia — Administration of conventional epidural analgesia using an 18G Tuohy needle for catheter placement and subsequent administration of a standardized dose of bupivacaine with fentanyl.
  Arms: Standard Epidural Analgesia
Procedure: Dural Puncture Epidural Analgesia — Administration of epidural analgesia that incorporates a dural puncture with a 27G spinal needle prior to epidural catheter placement, followed by the same standardized dose of bupivacaine with fentanyl.
  Arms: Dural Puncture Epidural (DPE) Analgesia

SUMMARY:
Childbirth is both a physically and emotionally intense experience for mothers. Today, epidural analgesia is used during labor to improve maternal comfort and help ensure a safe, controlled delivery. Standard epidural analgesia is one of the most common methods used; however, it can sometimes cause issues like a one-sided block, insufficient pain relief, or motor block.

In recent years, the dural puncture epidural (DPE) technique has emerged as an alternative method to enhance the effectiveness of epidural analgesia. In the DPE method, a 27G spinal needle is used to puncture the dura before placing the epidural catheter. This allows cerebrospinal fluid to be seen, but no medication is injected into the intrathecal space. It is believed that DPE improves the spread of the epidural medication, reduces the time needed for a sacral block, and creates a more even block.

The primary aim of this study is to compare the effectiveness of standard epidural analgesia and DPE during labor, by measuring the rate at which patients achieve adequate pain relief (NRS < 4).

The secondary aims are to compare both methods regarding:

Changes in blood pressure and heart rate during labor, Changes in fetal heart rate, Occurrence of motor block, Need for additional pain relief, Side effects (such as low blood pressure, itching, nausea, vomiting, and fetal bradycardia), Risk of post-dural puncture headache, and Patient satisfaction with pain management and overall childbirth experience. The results of this study will help determine which epidural technique is more effective and safe for use during labor, thus contributing to improved clinical practice.

DETAILED DESCRIPTION:
The process of childbirth is an intensely demanding experience for mothers, both physically and psychologically. Contemporary epidural analgesia techniques, employed during labor, not only enhance maternal comfort but also contribute to the safe and controlled progression of delivery. Although standard epidural analgesia is one of the most frequently preferred methods for labor pain management and provides effective pain control, it is sometimes associated with disadvantages such as unilateral block, inadequate analgesia, or motor block.

In recent years, the dural puncture epidural (DPE) technique has emerged as an alternative method to improve the efficacy of epidural analgesia. In the DPE method, the dura is punctured using a 27G spinal needle prior to the placement of the epidural catheter, allowing the observation of cerebrospinal fluid without the administration of intrathecal medication. It is postulated that the DPE technique enhances the spread of the epidural solution, shortens the time required to achieve sacral block, and yields a more homogeneous block.

The primary objective of this study is to compare the adequacy and effectiveness of standard epidural analgesia versus dural puncture epidural analgesia during labor. Adequacy will be evaluated by the proportion of patients achieving the target pain score (NRS < 4).

The secondary objectives include comparing the two techniques with respect to hemodynamic changes during labor, alterations in fetal heart rate, development of motor block, need for additional analgesia, incidence of side effects (such as hypotension, pruritus, nausea, vomiting, fetal bradycardia), and the risk of post-dural puncture headache. Additionally, the study will assess the impact of each method on patient satisfaction with both postoperative analgesia management and the overall childbirth experience.

The findings of this study aim to elucidate which epidural analgesia technique is more effective and safe for use during labor, thereby contributing to clinical practice improvements.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Gestational age of ≥36 weeks with vertex presentation
* In active labor with cervical dilation ≤5 cm
* Electing for a pain-free vaginal delivery with one of the two epidural analgesia methods
* Provision of written informed consent

Exclusion Criteria:

* Presence of pregnancy-related diseases (e.g., preeclampsia, gestational diabetes)
* Contraindications to neuraxial block
* Risk factors for cesarean delivery (e.g., uterine anomalies, previous surgeries, morbid obesity)
* Known fetal anomalies

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Adequate Analgesia Achievement (NRS < 4) | Assessed at 5, 10, and 15 minutes after each epidural dose administration.
  The primary outcome measure is the proportion of participants achieving a target pain score of less than 4 on the Numeric Rating Scale (NRS), a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicate worse pain, after each epidural dose administration. Additional doses, if required, will be administered as per protocol, with outcomes assessed following each dose.

SECONDARY OUTCOMES:
Maternal Hemodynamic Changes | Assessed every 10 minutes during labor.
  Variation in maternal blood pressure and heart rate during labor following each epidural dose administration.
Fetal Heart Rate Variations | Recorded every 10 minutes until delivery.
  Changes in fetal heart rate, monitored continuously during labor.
Incidence and Severity of Motor Block | From the first epidural dose until delivery completion (approximately 6 hours on average)
  Occurrence and degree of motor block, as evaluated by the Modified Bromage Scale-a scale ranging from 0 (no motor block) to 3 (complete motor block), where higher scores indicate more severe motor block-following each epidural dose.
Need for Additional Analgesia | From the first epidural dose until delivery, typically up to 12 hours
  Frequency of additional epidural dosing required for achieving adequate pain relief, defined as the administration of an extra dose when a Numeric Rating Scale (NRS) score of ≥ 4 is recorded (NRS: 0 [no pain] to 10 [worst possible pain], where higher scores indicate worse pain
Occurrence of Adverse Effects | Monitored at 10-minute intervals throughout labor.
  Recording of adverse effects including hypotension, pruritus, nausea, vomiting, and fetal bradycardia during labor.
Post-Dural Puncture Headache | up to 1 weeks
  Incidence and severity of post-dural puncture headache in the postpartum period.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication

REFERENCES:
- [Background] Lin W, Yang Y, Lin J, Chen J, Lin Q. Dural Puncture Epidural with 25-G Spinal Needles versus Conventional Epidural Technique in Conjunction with PIEB for Labor Analgesia: A Randomized Trial. J Pain Res. 2023 Nov 8;16:3797-3805. doi: 10.2147/JPR.S424082. eCollection 2023. PMID 38026464
- [Background] Song Y, Du W, Zhou S, Zhou Y, Yu Y, Xu Z, Liu Z. Effect of Dural Puncture Epidural Technique Combined With Programmed Intermittent Epidural Bolus on Labor Analgesia Onset and Maintenance: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):971-978. doi: 10.1213/ANE.0000000000004768. PMID 32282386
- [Background] Wang J, Zhang L, Zheng L, Xiao P, Wang Y, Zhang L, Zhou M. A randomized trial of the dural puncture epidural technique combined with programmed intermittent epidural boluses for labor analgesia. Ann Palliat Med. 2021 Jan;10(1):404-414. doi: 10.21037/apm-20-2281. PMID 33545772